CLINICAL TRIAL: NCT01392170
Title: Phase II Study of Pegylated Ifná-2a (Pegasys) in Patients With Chronic Myeloid Leukemia Who Have Minimal Residual Disease While Receiving Therapy With Tyrosine Kinase Inhibitors
Brief Title: Pegasys in Patients With Chronic Myeloid Leukemia (CML)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0184; NCI-2011-01465 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2015-04-14 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Leukemia
Keywords: Leukemia; Chronic Myeloid Leukemia; CML; Tyrosine Kinase Inhibitors; TKI; Complete cytogenetic remission; CCyR; Minimal residual disease; MRD; PEG-IFNa-2a; Pegasys; Peginterferon Alpha-2a; Philadelphia chromosome (Ph)-positive; BCR-ABL1-positive
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasm, Residual; Philadelphia Chromosome | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEG-IFNá-2a (Experimental): PEG-IFNá-2a (Pegasys) 45 mcg subcutaneously as single weekly dose.
  Interventions: Drug: PEG-IFNá-2a

INTERVENTIONS:
Drug: PEG-IFNá-2a — 45 mcg given subcutaneously as a single weekly dose for 24 months.
  Other Names: Pegasys; Peginterferon Alpha-2a

SUMMARY:
The goal of this clinical research study is to learn if adding pegylated interferon-alfa 2a (Pegasys) to the TKI that you are already receiving can help to control CML. The safety of this treatment combination will also be studied.

Pegasys is a form of the drug interferon. It is designed to help the body's immune system to fight infections. It may also affect the body's response to cancer.

A TKI (imatinib mesylate, nilotinib, or dasatinib) is designed to bind to and shut off a protein in tumor cells called Bcr-Abl. Shutting Bcr-Abl off may prevent CML cells from growing, and may cause them to die.

You are already receiving a TKI. This consent form will describe the administration of Pegasys, any tests and procedures that need to be performed while you are receiving Pegasys, and any risks/benefits there may be from receiving Pegasys.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive Pegasys through a needle under the skin 1 time each week while you are on study. You will be taught how to use the study drug at the first visit and will administer it to yourself at all future doses.

You will continue receiving the TKI you are already taking at the dose and frequency you have been receiving it when you began taking part in this study.

Study Visits:

At every study visit, you will be asked about any side effects you may have had and to list any drugs you may be taking.

Every 1-2 weeks for 8 weeks, then every 6-8 weeks after that, blood (about 1-2 teaspoons) will be drawn for routine tests.

Every 3 months for 6 months, then every 6-12 months after that, you will have a complete physical exam, including measurement of your vital signs.

Every 3-6 months for 1 year, you will have a bone marrow aspirate to check the status of the disease and to check for changes in your chromosomes.

Every 3-6 months for 1 year, then every 6-12 months after that, blood (about 1 teaspoon) will be drawn to check the levels of leukemia in the blood.

Length of Study:

You may continue taking Pegasys for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

This is an investigational study. Pegasys is FDA approved and commercially available for the treatment of CML. TKIs (imatinib, nilotinib, and dasatinib) are FDA approved and commercially available for the treatment of CML. The combination of these drugs to treat CML is investigational.

Up to 50 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 16 years or older with Philadelphia chromosome (Ph)-positive or BCR-ABL1-positive CML (as determined by cytogenetics, FISH, or PCR).
2. Patients are receiving an FDA-approved TKI for the management of CML.
3. Patients must have received TKI therapy for at least 24 months and not have increased their TKI dose in the last 6 months.
4. Patients must be in complete cytogenetic remission.
5. Patients must have detectable BCR-ABL1 transcript levels meeting at least one of the following criteria: 1. The patient has received therapy for at least 2 years and does not have a sustained major molecular response, or 2. The patient has received therapy for at least 5 years and does not have a sustained complete molecular response.
6. Patients must not have had a known continuous interruption of TKI therapy of greater than 14 consecutive days or for a total of 6 weeks in the 6 months prior to enrollment.
7. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study.
8. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
9. Adequate organ function defined as: bilirubin < 2x upper limit of normal (ULN) (unless associated with Gilbert's syndrome), creatinine </= 1.5x ULN, and serum glutamate pyruvate transaminase (sGPT) or serum glutamate oxaloacetate transaminase (sGOT) </= 2.5x ULN.
10. Men and women of childbearing potential should practice effective methods of contraception. Women of childbearing potential must have a negative serum or urine pregnancy test within 1 week of enrollment.

Exclusion Criteria:

1. Patients receiving any non-FDA approved TKI.
2. Patients who are pregnant or breast-feeding.
3. Patients with clinically significant heart disease (NYHA Class III or IV).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Quintas-Cardama, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 28, 2011 to March 28, 2013. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Study was terminated due to slow accrual.
Period: Overall Study
Arm/Group | PEG-IFNá-2a
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | PEG-IFNá-2a
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieved of Major Molecular Response (MMR) or Complete Molecular Response (CMR)
Description: Molecular response defined as: major molecular response (MMR) corresponds to a BCR-ABL1/ABL1 ratio of <=0.01. Complete molecular response (CMR) is defined as undetectable BCR-ABL1 transcripts. Molecular response measured every 3 months (a total of 4 assessments within one year of therapy).
Time Frame: 12 months from start of treatment with PEG-IFNá-2a
Population: Study terminated due to low accrual. No participants were evaluable for outcome.
Arm/Group | PEG-IFNá-2a
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection through 30 days post treatment.
Arm/Group | PEG-IFNá-2a
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Early termination due to slow accrual, no analysis possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes